CLINICAL TRIAL: NCT00380406
Title: PROtecting Ovaries and Fertility During Chemotherapy - The PROOF Trial: A Randomized Controlled Trial of Gonadotropin Releasing Hormone Agonist (GnRHa) for Fertility Preservation in Oncology Patients
Brief Title: PROtecting Ovaries and Fertility During Chemotherapy - The PROOF Trial
Acronym: PROOF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: University of Ottawa (Other); Queen's University (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006603-01H
Record Dates: First submitted 2006-09-23; First posted 2006-09-26 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2010-08

CONDITIONS: Fertility Preservation; Cancer
Keywords: Gonadotropin releasing hormone agonist; GnRH; Fertility; Fertility preservation; Oncology; Cancer; Chemotherapy
MeSH Terms: conditions — Neoplasms | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Leuprolide acetate
- depot GnRHa (Leuprolide acetate (LA) 11.25 mg intramuscularly) (Active Comparator)
  Interventions: Drug: Leuprolide acetate

INTERVENTIONS:
Drug: Leuprolide acetate

SUMMARY:
The purpose of this study is to determine whether gonadotropin releasing hormone agonists (medical therapy) will protect against ovarian failure in reproductive aged women undergoing sterilizing chemotherapy.

DETAILED DESCRIPTION:
Fertility preservation is defined as the maintenance of one's ability to reproduce.

The hypothesis for this study is that medical treatment (GnRHa) will help female cancer patients, receiving sterilizing chemotherapy, preserve their ovarian function and therefore fertility. This study is a feasibility trial of the drug (GnRHa)vs placebo in female cancer patients receiving gonadotoxic chemotherapy between the ages of 18 and 38 who wish to participate.

The objective of the feasibility trial is to determine the feasibility of a definitive study to answer this question and also to define the required parameters needed to design the definitive study such as the observable difference in ovarian failure between the drug and placebo groups. The same protocol will be followed as proposed for the definitive trial but with a smaller sample size.

This pilot study will be conducted at the Ottawa Hospital Regional Cancer Centre/Division of Reproductive Medicine of Department of Obstetrics and Gynecology, University of Ottawa and the Cancer Centre of Southeastern Ontario/Division of Reproductive Medicine of Department of Obstetrics and Gynecology, University of Ottawa.

The planned trial intervention is trimonthly (every 3 months) administration of depot GnRHa (Leuprolide acetate (LA) 11.25 mg intramuscularly) or placebo. Injections would start prior to initiation of chemotherapy, in the luteal phase of the menstrual cycle preceding chemotherapy, and will continue until cessation of chemotherapy (maximum of 6 months or 2 injections). Since only adjuvant/curative chemotherapy patients will be enrolled, chemotherapy will last a maximum of six months.

Subjects will be randomized, with concealed allocation, to either GnRHa or placebo. Subjects and investigators will be blinded to the intervention administered.

Inclusion criteria: Women who are

1. between ages 18 to 38;
2. who will be undergoing gonadotoxic (sterilizing) curative/ adjuvant chemotherapy for early stage disease; and
3. have provided informed consent. All subjects will be enrolled from the Ottawa Hospital Regional Cancer Institute (OHRCC) and the Cancer Center of South Eastern Ontario at Kingston General Hospital (CCSEO). Gonadotoxic chemotherapy includes alkylating / anthracycline agents eg. cyclophosphamide.

Exclusion criteria: Women who;

1. have advanced stage disease and/or whose median survival is expected to be less than 6 months
2. have cancer of the ovaries, uterus, or fallopian tubes;
3. have clinical or biochemical evidence of diminished ovarian reserve (recent shortening of cycles < 24 days between menses, age > 38, elevated serum FSH (follicular stimulating hormone)> 15 IU/L, or low antral follicle count (AFC- number of follicles less than 10 mm on day 2 or 3 of natural menses) on baseline pelvic ultrasound (<5) or elevated day 2 or 3 estradiol (> 280 pmol/ml);
4. have previously received chemotherapy or abdominal/pelvic radiation or have planned to receive abdomino/pelvic radiation;
5. are pregnant;
6. have contraindications to intramuscular injections; or 7) have a history of fractures secondary to/or documented osteoporosis.

Outcomes: Subjects will be assessed at baseline, monthly (for adverse effects only) during active intervention, and at 0, 3, 6, 9, and 12 months post cessation of chemotherapy and treatment (GnRHa/ placebo) for predictors of ovarian reserve.

The primary outcome is protection against ovarian failure at 12 months post chemotherapy. This is measured by resumption of regular menstrual cycles (every 24 -35 days) with documentation of ovulation by biochemistry (progesterone levels) over a minimum of three months.

Secondary outcomes will include sonographic (biophysical) and biochemical markers of ovarian reserve.

ELIGIBILITY:
Inclusion Criteria:

* Women who are:

  1. between ages 18 to 38;
  2. who will be undergoing gonadotoxic (sterilizing) curative/ adjuvant chemotherapy for early stage disease; and
  3. have provided informed consent. All subjects will be enrolled from the Ottawa Hospital Regional Cancer Institute (OHRCC) and the Cancer Center of South Eastern Ontario at Kingston General Hospital (CCSEO).

Exclusion Criteria:

* Women who:

  1. have advanced stage disease and/or whose median survival is expected to be less than 6 months
  2. have cancer of the ovaries, uterus, or fallopian tubes;
  3. have clinical or biochemical evidence of diminished ovarian reserve (recent shortening of cycles < 24 days between menses, age > 38, elevated serum FSH (follicular stimulating hormone)> 15 IU/L, or low antral follicle count (AFC- number of follicles less than 10 mm on day 2 or 3 of natural menses) on baseline pelvic ultrasound (<5) or elevated day 2 or 3 estradiol (> 280 pmol/ml);
  4. have previously received chemotherapy or abdominal/pelvic radiation or have planned to receive abdomino/pelvic radiation;
  5. are pregnant;
  6. have contraindications to intramuscular injections; or
  7. have a history of fractures secondary to/or documented osteoporosis.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-01; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Protection against ovarian failure | 12 months post Chemo therapy

SECONDARY OUTCOMES:
Sonographic (biophysical) and biochemical markers of ovarian reserve | 3,6,9,12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sonya Kashyap, MD MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (4):
- Canada (4):
  - Cancer Centre of Southeastern Ontario, Kingston, Ontario
  - Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Kingston General Hospital, Ottawa, Ontario
  - Ottawa Hospital/OHRI, Ottawa, Ontario